CLINICAL TRIAL: NCT04082637
Title: Mindful Body Awareness Training as an Adjunct to Medication Treatment for Opioid Use Disorder
Brief Title: Mindful Body Awareness With Medication Treatment for Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Cynthia Price, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00005923; R33AT009932 (NIH); R21AT009932 (NIH); R01AT010742 (NIH)
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Opioid-use Disorder
Keywords: Buprenorphine; Medication-assisted treatment; Mind-body therapies; Mindfulness; Interoception; Mindful Awareness in Body-oriented Therapy
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MABT* + Medication Treatment (Experimental): Mindful Awareness in Body-oriented Therapy + Medication Treatment
  Interventions: Behavioral: Mindful Awareness in Body-oriented Therapy
- Treatment as Usual (No Intervention): Treatment as Usual is medication for the treatment of opioid use disorder

INTERVENTIONS:
Behavioral: Mindful Awareness in Body-oriented Therapy — A mind-body intervention designed to teach interoceptive awareness skills for emotion regulation and self-care. Delivered individually in 75 minute sessions once a week for 8 weeks.
  Other Names: MABT
  Arms: MABT* + Medication Treatment

SUMMARY:
The national opioid epidemic requires development of real-world evidence-based treatments for opioid use disorder, including adjuncts to Medication for Opioid Use Disorder (MOUD). Interventions are needed that address the complex needs of patients with opioid use disorder, which include substantial mental health co-morbidity and high rates of chronic pain related to the complex interaction of opioid prescribing for pain and opioid use disorder. This study leverages recent federal and state opioid use disorder treatment initiatives as a platform for testing a promising mind-body intervention, Mindful Awareness in Body-oriented Therapy (MABT) as an adjunct to MOUD in multiple clinical settings funded primarily through the Washington Opioid State Targeted Response (STR) program. MABT, a novel mindfulness-based intervention, uniquely addresses aspects of awareness, interoception, and regulation that may be associated with pain, mental health distress, and behavioral control that increase risk of relapse and poor treatment outcomes. Using a randomized, two-group, repeated measures design, we will compare those who receive MABT+ MOUD vs. MOUD only. The overarching goal of this application is to test MABT to improve MOUD health outcomes. The specific aims for the combined R33/R01 clinical protocol are to: 1) evaluate the effectiveness of MABT + TAU (MOUD) compared to TAU only in reducing opioid use and other substances; 2) examine the effectiveness of MABT + TAU to improve mental and physical health vs. TAU only; 3) examine the effectiveness of MABT + TAU to positively affect substance use related outcomes of craving and treatment retention vs. TAU only. For the R01, there is an additional aim to explore the effectiveness of additional MABT dose offered at 6 months to those with continued substance use (non-responders) compared to those with continued substance use at 6 months in TAU. A two-group (n = 165/165), randomized controlled repeated measures design will be employed. Three hundred thirty individuals engaged in MOUD will be recruited for participation at outpatient treatment sites. Assessments will be administered at baseline, post-intervention (3 months from baseline), and at 6, 9, and 12 months. Results of this study will inform the evidence base for behavioral treatment adjuncts to MOUD and directly impact the future direction of the Washington Opioid STR program.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with opioid use disorder
* enrolled in a medication treatment program for opioid use disorder
* is stable in program involving, (if on buprenorphine) Rx appointments less frequent than once/week; (if on methadone) at least 90 days in treatment with a minimum dose of 60mg, no missed dose evaluation appointments in past 30 days, and no more than 3 missed doses in 30 days
* willing to forego (non-study) manual (e.g., massage) and/or mind-body therapies (e.g., mindfulness meditation) for 3 months
* willing to sign release for access of electronic medical records
* fluent in English
* able to attend study sessions when offered

Exclusion Criteria:

* unwilling or unable to remain in MT treatment for the duration of the trial (includes planned relocation, pending incarceration, planned surgical procedures, etc.)
* over 24 weeks gestation or unknown gestation, if pregnant
* reports, or is noted by clinical or study staff as showing, overt psychosis or other conditions such as cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Time Line Follow-back | 90 days
  Patient-reported days of opioid use and other substances

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Price, PhD, Principal Investigator — University of Washington
Locations (5):
- United States (5):
  - Cascade Medical Advantage, Bellingham, Washington
  - North Olympic Health Network, Port Angeles, Washington
  - Harborview Hospital, Seattle, Washington
  - Country Doctors Clinics, Seattle, Washington
  - Evergreen Treatment Services, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Please see link below to access shared data, housed with ICPSR
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: currently available with no time limit
Access Criteria: apply to ICPSR for access
URL: http://doi.org/10.3886/ICPSR39235

REFERENCES:
- [Result] Price CJ, Merrill JO, McCarty RL, Pike KC, Tsui JI. A pilot study of mindful body awareness training as an adjunct to office-based medication treatment of opioid use disorder. J Subst Abuse Treat. 2020 Jan;108:123-128. doi: 10.1016/j.jsat.2019.05.013. Epub 2019 May 23. PMID 31174929
- [Result] Leyde S, Price CJ, Colgan DD, Pike KC, Tsui JI, Merrill JO. Mental Health Distress Is Associated With Higher Pain Interference in Patients With Opioid Use Disorder Stabilized on Buprenorphine or Methadone. Subst Use Addctn J. 2024 Jul;45(3):423-433. doi: 10.1177/29767342241227402. Epub 2024 Feb 7. PMID 38327009
- [Result] Rodriguez MN, Colgan DD, Leyde S, Pike K, Merrill JO, Price CJ. Trauma exposure across the lifespan among individuals engaged in treatment with medication for opioid use disorder: differences by gender, PTSD status, and chronic pain. Subst Abuse Treat Prev Policy. 2024 May 3;19(1):25. doi: 10.1186/s13011-024-00608-8. PMID 38702783
- [Result] Price CJ, Pike KC, Treadway A, Palmer JK, Merrill JO. Immediate Effects of Mindful Awareness in Body-Oriented Therapy as an Adjunct to Medication for Opioid Use Disorder. Mindfulness (N Y). 2024 Nov;15(11):2794-2811. doi: 10.1007/s12671-024-02463-x. Epub 2024 Nov 19. PMID 39697819
- [Derived] Price CJ, Pike KC, Merrill JO. Longitudinal effects of interoceptive awareness training as an adjunct to medication treatment for opioid use disorder: A randomized clinical trial of Mindful Awareness in Body-oriented Therapy. Drug Alcohol Depend. 2025 Oct 1;275:112813. doi: 10.1016/j.drugalcdep.2025.112813. Epub 2025 Aug 5. PMID 40784065
- [Derived] Price CU, Pike KC, Treadway A, Palmer J, Merrill JO. Immediate Effects of Mindful Awareness in Body-oriented Therapy as an Adjunct to Medication for Opioid Use Disorder. Res Sq [Preprint]. 2024 Jul 15:rs.3.rs-4727162. doi: 10.21203/rs.3.rs-4727162/v1. PMID 39070653
- [Derived] Rodriguez MN, Colgan DD, Leyde S, Pike K, Merrill JO, Price CJ. Trauma Exposure Across the Lifespan among Individuals Engaged in Treatment with Medication for Opioid Use Disorder: Differences by Gender, PTSD Status, and Chronic Pain. Res Sq [Preprint]. 2023 Dec 19:rs.3.rs-3750143. doi: 10.21203/rs.3.rs-3750143/v1. PMID 38196650

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT04082637/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT04082637/ICF_000.pdf